CLINICAL TRIAL: NCT03076502
Title: The Role of ctDNA, PVT1 and ROS in Diagnosis and Treatment of Gastrointestinal and Hepatobiliary Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Changzheng Hospital (Other); The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: ctDNA-GI
Record Dates: First submitted 2017-03-05; First posted 2017-03-10 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Neoplasms, Gastrointestinal
Keywords: ctDNA; Gastrointestinal Cancer; ROS; Hepatobiliary Pancreatic Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples; Portal vein blood samples; Tumor tissue samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the role of ct-DNA, PVT1 and reactive oxygen species (ROS) as biomarkers in the diagnosis, treatment and recurrence monitoring of gastrointestinal and hepatobiliary pancreatic cancer.

DETAILED DESCRIPTION:
Epidemiological surveys showed a significant increasing trend of gastrointestinal and hepatobiliary pancreatic cancer in recent years. How can make an early diagnosis of gastrointestinal and liver cancer as well as prognostic evaluation and efficacy monitoring, has become the hotspot. "liquid biopsy", which is meant to detect cancers by sequencing the DNA in a few drops of a person's blood. It may detect cancers early, even before symptoms arise, when there is just a few cells in the blood circulation.

ct-DNA in cancer patients often bears similar genetic and epigenetic features to the related tumor DNA. There is evidence that some of the ct-DNA originates from tumoral tissue. Besides, ct-DNA can easily be isolated from the circulation and other body fluids of patients, makes it a promising candidate as a non-invasive biomarker of cancer.

It is known that levels of cellular ROS correlate with the aggressiveness of tumour cells and prognosis of patients. Cancer cells with increased endogenous ROS stress are more sensitive to anticancer agents and high levels of ROS generated by chemotherapeutic agents can induce cell death. Hence, ROS levels before and after chemotherapy in cancer cells can be an early indicator of treatment efficacy, which has the potential to shed new light on the choice of cancer therapy.

This study aims to evaluate the role of ct-DNA and ROS as biomarkers in the diagnosis, treatment and recurrence monitoring of gastrointestinal and hepatobiliary pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected of gastrointestinal and hepatobiliary pancreatic cancer
* Age from 18 - 80 years
* No serious organic and mental illness;

Exclusion Criteria:

* Pregnancy
* No pathologic result
* Suffering other malignancies at the same time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected gastrointestinal and hepatobiliary pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Pathological diagnosis | intraoperative
  Sensitivity and specificity

SECONDARY OUTCOMES:
Tumor status（worse/ maintain/ better） | 2 years
  the level of ct-DNA compared with the tumor burden

CONTACTS AND LOCATIONS:
Overall Officials: JIAN WANG, M.D., Principal Investigator — Department of Biliary-pancreatic Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: No